CLINICAL TRIAL: NCT03427814
Title: A Phase 2, Double-blind, Randomized Study of BGB-290 Versus Placebo as Maintenance Therapy in Patients With Inoperable Locally Advanced or Metastatic Gastric Cancer That Responded to Platinum-based First-line Chemotherapy
Brief Title: Study of BGB-290 or Placebo in Participants With Advanced or Inoperable Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-290-303; 2017-003493-13 (EudraCT Number); CTR20171664 (Registry Identifier: Center for drug evaluation NMPA)
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Advanced or Inoperable Gastric Cancer
Keywords: BGB-290; PARP inhibitor; Phase 2; maintenance therapy; gastric cancer; oral treatment; PARALLEL 303; PARALLEL; BGB290303; BGB-290-303
MeSH Terms: conditions — Stomach Neoplasms | interventions — pamiparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pamiparib (Experimental): Participants received pamiparib orally.
  Interventions: Drug: Pamiparib
- Placebo (Placebo Comparator): Participants received placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pamiparib — 60 mg orally twice daily
  Other Names: BGB-290
  Arms: Pamiparib
Drug: Placebo — 60 mg orally twice daily
  Arms: Placebo

SUMMARY:
This study enrolled participants with previously-treated advanced or inoperable gastric cancer who have responded to first line platinum therapy into two treatment arms. In Arm A participants received BGB-290; in Arm B participants received placebo. The purpose of this study is to show that BGB-290 (pamiparib) (versus placebo) will improve progression-free survival (PFS) in participants with advanced or inoperable gastric cancer.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled, randomized multicenter global phase 2 study comparing the efficacy and safety of single agent poly (ADP-ribose) polymerase (PARP) inhibitor BGB-290 to placebo as maintenance therapy in participants with advanced gastric cancer who have responded to first line platinum based chemotherapy. Participants are randomized 1:1 to BGB-290 (Arm A) or placebo (Arm B). Randomization will be stratified by geography, biomarker status, and ECOG performance status.

Participants will undergo tumor assessments at screening and then every 8 weeks, or as clinically indicated. Administration of BGB-290 or placebo will continue until disease progression, unacceptable toxicity, death, or another discontinuation criterion is met.

After end of treatment, long-term follow-up assessments include tumor imaging every 8 weeks for those participants without disease progression, survival status, and new anticancer therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years.
2. Signed informed consent.
3. Histologically confirmed inoperable locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction.
4. Received platinum based first line chemotherapy for ≤ 28 weeks.
5. Confirmed partial response (PR) maintained for ≥ 4 weeks or complete response (CR).
6. Able to be randomized to study ≤ 8 weeks after last platinum dose.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
8. Adequate hematologic, renal and hepatic function.
9. Must be able to provide archival tumor tissue for central biomarker assessment.
10. Females of childbearing potential and non-sterile males must agree to use highly effective methods of birth control throughout the course of study and at least up to 6 months after last dosing.

Key Exclusion Criteria:

1. Unresolved acute effects of prior therapy ≥ Grade 2.
2. Prior treatment with PARP inhibitor.
3. Chemotherapy, biologic therapy, immunotherapy or other anticancer therapy ≤ 14 days prior to randomization.
4. Major surgery or significant injury ≤ 2 weeks prior to start of study treatment.
5. Diagnosis of myelodysplastic syndrome (MDS)
6. Other diagnoses of significant malignancy
7. Leptomeningeal disease or brain metastasis
8. Inability to swallow capsules or disease affecting gastrointestinal function.
9. Active infections requiring systemic treatment.
10. Clinically significant cardiovascular disease
11. Pregnant or nursing females.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (65):
- United States (7):
  - Miami Cancer Institute, Miami, Florida
  - Scri Florida Cancer Specialist East, West Palm Beach, Florida
  - Goshen Center For Cancer Care, Goshen, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Novant Health Hematology Charlotte, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
- Australia (4):
  - Gosford Hospital, Gosford, New South Wales
  - Monash Health, Clayton, Victoria
  - Ballarat Oncology and Haematology Services, Wendouree, Victoria
  - St John of God Health Care, Subiaco, Western Australia
- Belgium (2):
  - Az Sint Jan Brugge, Bruges
  - University Hospitals Leuven, Leuven
- China (10):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
- Fakultni Nemocnice Bulovka, Prague, Czechia
- France (9):
  - Chru de Brest Hospital Morvan, Brest
  - Chu Besancon Hopital Jean Minjoz, Doubs
  - Hopital Prive Jean Mermoz, Lyon
  - Icm Val Daurelle Oncologie Medicale, Montpellier
  - Hopital Prive Des Cotes Darmor Service Oncologie, Plérin
  - Centre Eugene Marquis, Rennes
  - Ico Site Rene Gauducheau, SaintHerblain
  - Iuc Toulouse Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Acad Fridon Todua Medical Center Ltd Research Institute of Clinical Medicine Ltd, Tbilisi, Georgia
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (2):
  - Orszagos Onkologiai Intezet, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Japan (7):
  - Nho Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kindai University Nara Hospital, Ikoma, Nara
  - Oita University Hospital, Yufushi, Oita Prefecture
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suitashi, Osaka
  - Saitama Medical University International Medical Center, Hidakashi, Saitama
  - Showa University Koto Toyosu Hospital Oncology, Koto, Tokyo
- Poland (4):
  - Szpitale Pomorskie Spolka Z Ograniczona Odpowiedzialnoscia, Gdynia
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw
  - Mazowiecki Szpital Onkologiczny, Wieliszew
- Russia (5):
  - Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Regional Buz Kurskiy Regional Clinical Oncologic Dispensary, Kursk, Kursk Oblast
  - Bih of Omsk Region Clinical Oncology Dispensary, Omsk, Omsk Oblast
  - Pavlov First Saint Petersburg State Medical University, SaintPetersburg, Sankt-Peterburg
  - State Budgetary Healthcare Institution Volgograd Regional Clinical Oncology Dispensary, Volgograd, Volgograd Oblast
- Tan Tock Seng Hospital Oncology, Singapore, Singapore
- Spain (8):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall Dhebron, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Clinica Universidad de Navarra Pamplona, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia
- Chi Mei Medical Center, Tainan, Taiwan
- United Kingdom (2):
  - Sarah Cannon Research Institute Uk, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in Asia, Australia, Europe, and North America.
Groups:
- Pamiparib: Participants received 60 milligrams (mg) pamiparib orally twice a day until progressive disease, unacceptable toxicity, death, or withdrawal of consent for study treatment, investigator's discretion, start of new anticancer therapy or Sponsor's decision to end the study
- Placebo: Participants received 60 mg placebo orally twice daily until progressive disease, unacceptable toxicity, death, withdrawal of consent for study treatment, investigator's discretion, start of new anticancer therapy, or Sponsor's decision to end the study
Period: Overall Study
Arm/Group | Pamiparib | Placebo
Started | 71 | 65
Completed | 0 | 0
Not Completed | 71 | 65
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 42 | 31
Not completed — Sponsor's Decision | 1 | 0
Not completed — Investigator's Decision | 1 | 2
Not completed — Disease progression | 1 | 0
Not completed — Treatment Completed | 0 | 1
Not completed — Sponsor's Decision to End study | 21 | 25
Not completed — Transfer to Long Term Extension Study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Analysis Set included all randomized participants who were assigned to a study drug (pamiparib or placebo)
Groups:
- Pamiparib: Participants received 60 mg pamiparib orally twice a day until progressive disease, unacceptable toxicity, death, or withdrawal of consent for study treatment, investigator's discretion, start of new anticancer therapy or Sponsor's decision to end the study
- Total: Total of all reporting groups
Arm/Group | Pamiparib | Placebo | Total
Number analyzed (Participants) | 71 | 65 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.82) | 62.1 (11.23) | 62.3 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 46 | 45 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 53 | 50 | 103
  Unknown or Not Reported | 14 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 15 | 35
  Black or African America | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 38 | 36 | 74
  Other | 1 | 3 | 4
  Not Reported/Unknown | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Investigator Assessment
Description: PFS is defined as the time from randomization to progressive disease (PD) per Response Evaluation Criteria in Solid Tumors ( RECIST) Version 1.1 by investigator assessment or death due to any cause, whichever occurs first.
Time Frame: Approximately 23 months
Population: Intent To Treat (ITT) Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 71 | 65
Months | 3.7 [1.94 to 5.26] | 2.1 [1.87 to 3.75]
Statistical Analysis 1: Comparison: Pamiparib vs Placebo; Test type: Superiority; p = 0.1428, Log Rank; The one-sided p-value was based on a stratified log-rank test

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Approximately 23 months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 71 | 65
Months | 10.2 [8.71 to 16.33] | 12.0 [8.21 to NA] — NA = Not Estimable due to insufficient number of events

3. Secondary Outcome: Time To Second Subsequent Treatment (TSST)
Description: TSST is defined as the time from randomization until the second subsequent anticancer therapy or death after next-line therapy
Time Frame: Approximately 23 months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 71 | 65
Months | 9.8 [8.05 to 10.94] | 9.7 [7.49 to 14.00]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of Complete Response or Partial Response per RECIST Version 1.1 by investigator assessment
Time Frame: Approximately 23 months
Population: Efficacy Evaluable Analysis Set includes all randomized participants who had measurable disease at baseline and had at least one post baseline tumor assessment unless discontinued treatment due to clinical progression or death prior to tumor assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 39 | 32
Percentage of participants | 7.7 [1.62 to 20.87] | 6.3 [0.77 to 20.81]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first documented confirmed response of Complete Response or Partial Response to progressive disease (PD) per RECIST Version 1.1 by investigator assessment or death due to any cause, whichever occurs first
Time Frame: Approximately 23 months
Population: Efficacy Evaluable Analysis Set; Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 3 | 2
Months | 3.6 [3.48 to NA] — NA = Not estimable due to insufficient number of events | NA [5.55 to NA] — NA = Not estimable due to insufficient number of events

6. Secondary Outcome: Time To Response
Description: Time to response is defined as the time from randomization to the first documented response of Complete Response or Partial Response per RECIST Version 1.1 by investigator assessment
Time Frame: Approximately 23 months
Population: Efficacy Evaluable Analysis Set; Only responders were included in the analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 3 | 2
Months | 3.68 [1.8 to 7.3] | 1.87 [1.87 to 1.9]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From start of study treatment until 30 days after the last study drug intake or initiation of new anticancer therapy, whichever occurs first (up to approximately 4 years and 5.5 months)
Population: Safety Analysis Set includes all participants in the ITT Analysis Set who receive at least one dose of study treatment (pamiparib or placebo).
Measure: Number; unit: Number of participants
Arm/Group | Pamiparib | Placebo
Number analyzed (Participants) | 71 | 65
Number of participants
  Participants With At Least 1 TEAE | 66 | 61
  Participants with Serious TEAEs | 17 | 11

ADVERSE EVENTS:
Time Frame: From start of study treatment until 30 days after the last study drug intake or initiation of new anticancer therapy, whichever occurs first (up to approximately 4 years and 5.5 months)
Description: Safety Analysis Set includes all participants in the ITT Analysis Set who receive at least one dose of study treatment (pamiparib or placebo).
Arm/Group | Pamiparib | Placebo
All-Cause Mortality (participants affected / at risk) | 42/71 | 31/65
Serious Adverse Events (participants affected / at risk) | 17/71 | 11/65
Other Adverse Events (participants affected / at risk) | 65/71 | 57/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pamiparib (N=71) | Placebo (N=65)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malignant dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hepatic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pamiparib (N=71) | Placebo (N=65)
Anaemia (Blood and lymphatic system disorders) | 25 (31) | 10 (12)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (8) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (7) | 5 (7)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 13 (14)
Abdominal pain upper (Gastrointestinal disorders) | 12 (13) | 7 (7)
Constipation (Gastrointestinal disorders) | 9 (13) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 13 (21) | 9 (10)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 7 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 23 (26) | 12 (14)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 16 (17) | 2 (2)
Asthenia (General disorders) | 16 (16) | 12 (12)
Chest pain (General disorders) | 3 (5) | 0 (0)
Fatigue (General disorders) | 4 (4) | 4 (4)
Malaise (General disorders) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 6 (6) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (3)
Alanine aminotransferase increased (Investigations) | 8 (9) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 9 (11) | 5 (6)
Blood alkaline phosphatase increased (Investigations) | 6 (6) | 4 (6)
Blood bilirubin increased (Investigations) | 3 (4) | 1 (2)
Blood creatinine increased (Investigations) | 5 (5) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 3 (3)
Lymphocyte count decreased (Investigations) | 4 (4) | 1 (3)
Neutrophil count decreased (Investigations) | 7 (17) | 3 (4)
Platelet count decreased (Investigations) | 8 (10) | 2 (3)
Weight decreased (Investigations) | 9 (9) | 2 (2)
Weight increased (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 8 (16) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 19 (21) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (2) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 9 (10)
Insomnia (Psychiatric disorders) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (3) | 2 (3)
Hypotension (Vascular disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03427814/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT03427814/SAP_001.pdf